CLINICAL TRIAL: NCT03600038
Title: Pilot Trial of a Smartphone Smoking Cessation Application Intervention for Cancer Patients (Quit2Heal Study)
Brief Title: Smoking Cessation Smartphone App for Cancer Patients (Quit2Heal Study)
Acronym: Quit2Heal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); CVS Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8630; NCI-2018-02641 (Registry Identifier: NCI / CTRP); RG1001682 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Cancer; Smoking
Keywords: Smoking cessation; App for quitting smoking; Cancer; Oncology
MeSH Terms: conditions — Neoplasms; Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This is the experimental arm of the study. This includes receiving the novel/experimental smoking cessation smartphone app. Therapy description of experimental app withheld to protect the integrity of the study.
  Interventions: Behavioral: Experimental smoking cessation smartphone app
- Control (Active Comparator): This is the control arm of the study. This includes receiving the standard of care smoking cessation smartphone app. Therapy description of standard of care app withheld to protect the integrity of the study.
  Interventions: Behavioral: Standard of care smoking cessation smartphone app

INTERVENTIONS:
Behavioral: Experimental smoking cessation smartphone app — The experimental arm includes an intervention using a novel/experimental smartphone smoking cessation app.
  Arms: Experimental
Behavioral: Standard of care smoking cessation smartphone app — The control intervention uses a standard of care smartphone smoking cessation app.
  Arms: Control

SUMMARY:
The goal of this study is to determine whether the novel smartphone application designed specifically for cancer patients to quit smoking (Quit2Heal) provides higher quit rates than the current standard smoking cessation app.

DETAILED DESCRIPTION:
Cigarette smoking has harmful effects on cancer patients' treatment and prognosis, but there are systemic barriers to delivering smoking cessation interventions to cancer patients. One solution for addressing these barriers is to give patients immediate access to smoking cessation treatment via a smartphone application. The Quit2Heal smartphone app is engaging and tailored to the specific needs of cancer patients, and can be integrated into routine cancer care. The goal of this study is to determine whether Quit2Heal provides higher quit rates than the current standard smoking cessation app.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* diagnosed with cancer in the past 12 months
* has smoked a cigarette (even a puff) in the past 30 days
* interested in learning skills to quit smoking
* willing to be randomly assigned to either smartphone application
* resides in US
* has at least daily access to their own smartphone
* knows how to login and download a smartphone application from the Apple app store or Android Play app store
* willing and able to read in English
* not currently using cessation medications or enrolled in other smoking cessation programs, and
* has never used the NCI's Quit Guide smartphone application.
* willing and able to complete one follow-up survey
* willing to provide email, phone, and mailing address.

Exclusion Criteria:

* The exclusion criteria are opposite of the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
30-day point prevalence abstinence | 2 months post randomization
  No smoking in the past 30 days, as reported 2 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bricker JB, Watson NL, Heffner JL, Sullivan B, Mull K, Kwon D, Westmaas JL, Ostroff J. A Smartphone App Designed to Help Cancer Patients Stop Smoking: Results From a Pilot Randomized Trial on Feasibility, Acceptability, and Effectiveness. JMIR Form Res. 2020 Jan 17;4(1):e16652. doi: 10.2196/16652. PMID 31951215
- See also: Quit2Heal Study recruitment website — http://www.quit2heal.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03600038/Prot_SAP_000.pdf